CLINICAL TRIAL: NCT01843322
Title: Endoleak Repair Guided by Navigation Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: SINTEF Health Research (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011/720
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Aortic Aneurysm; Endoleak
Keywords: Image guided therapy; Endovascular procedures; Angiography; Vascular surgical procedures
MeSH Terms: conditions — Aortic Aneurysm; Endoleak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- navigation technology (Experimental): custom made navigation technology integrated in a Siemens angiography suite for feasibility evaluation in endoleak repair procedure
  Interventions: Procedure: endoleak repair procedure (navigation technology )

INTERVENTIONS:
Procedure: endoleak repair procedure (navigation technology )

SUMMARY:
The study is aimed at investigating whether repair of endoleak type II can be improved by adding navigation technology. Can this technology increase precision by guiding the needle that punctures through the skin as used during the repair procedure? Can the procedure logistics be improved by using navigation technology instead of computed tomography (CT) guidance of the needle puncture? Parameters logged during the procedure:

* was the needle placement successful?
* number of needle punctures?
* time used on guidance procedure
* X-ray exposure dose

ELIGIBILITY:
Inclusion Criteria:

* detected endoleak

Exclusion Criteria:

* n/a

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
detected leakage | within 1 hour after intervention
  number of patients with persistent leakage

CONTACTS AND LOCATIONS:
Overall Officials: Petter Aadahl, MD Prof, Study Director — National Taiwan Normal University
Locations (1):
- St Olavs Hospital, Trondheim, Norway